CLINICAL TRIAL: NCT05538520
Title: Effects of Stretching in a Conditioning Program Based on Pilates Exercises on Flexibility, Strength, Power and Muscular Endurance
Brief Title: Effects of Pilates Stretching on Flexibility, Strength, Power and Muscular Endurance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Estadual do Norte do Parana (Other)
Responsible Party: Principal Investigator, Raphael Goncalves de Oliveira, Professor, Universidade Estadual do Norte do Parana
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Pilates_stretching
Record Dates: First submitted 2022-09-06; First posted 2022-09-14 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-08

CONDITIONS: Young Adults; Performance; Exercise
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: Randomized and controlled clinical trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional Pilates (Experimental): 5 stretching exercises will be performed, followed by 15 strengthening exercises (5 for core, 5 for lower limbs and 5 for upper limbs), all in a series of 10 repetitions, 3x-week, for 8 weeks, maintaining an effort level 7-8 on the Omni-Scale. Below are the exercises and equipment used.
  1) Stretching the Chain Posterior (Reformer); 2) Front Splits Modified (Reformer); 3) Stomach Massage (Reformer); 4) Stretches Front (Barrel); 5) Back Stretches: Quadriceps Stretch (Barrel); 6) Bridge (Mat with Magic Circle); 7) The Hundred (Mat with Swiss ball); 8) Teaser (Mini Barrel); 9) Swan (Mini Barrel); 10) Swimming (Mini Barrel); 11) Footwork Double Leg Pumps (Chair); 12) Pump One Leg Front (Chair); 13) Forward Lunge (Chair); 14) Wall Side (Wall with Swiss ball and dumbbells); 15) Tower (Cadillac); 16) Arms Pulling Up (Cadillac); 17) Rowing Front: Hug a Tree (Cadillac); 18) Arm Pulling Down (Wall Unit); 19) Horizontal Arm Pulling (Wall Unit); 20) Extension Arm Up (Wall Unit).
  Interventions: Other: Traditional Pilates
- Pilates without stretching (Experimental): 15 strengthening exercises will be performed (the same performed by the TP group), all in a series of 10 repetitions, 3x-week, for 8 weeks, maintaining an effort level 7-8 on the Omni-Scale. Below are the exercises and equipment used.
  1) Bridge (Mat with Magic Circle); 2) The Hundred (Mat with Swiss ball); 3) Teaser (Mini Barrel); 4) Swan (Mini Barrel); 5) Swimming (Mini Barrel); 6) Footwork Double Leg Pumps (Chair); 7) Pump One Leg Front (Chair); 8) Forward Lunge (Chair); 9) Wall Side (Wall with Swiss ball and dumbbells); 10) Tower (Cadillac); 11) Arms Pulling Up (Cadillac); 12) Rowing Front: Hug a Tree (Cadillac); 13) Arm Pulling Down (Wall Unit); 14) Horizontal Arm Pulling (Wall Unit); 15) Extension Arm Up (Wall Unit).
  Interventions: Other: Pilates without stretching

INTERVENTIONS:
Other: Traditional Pilates — This group will perform a traditional Pilates session, which consists of stretching exercises, followed by exercises to strengthen the core (trunk flexors and extensors), lower limbs and upper limbs. The total duration of the intervention in this group should be approximately 50 minutes.
  Arms: Traditional Pilates
Other: Pilates without stretching — This group will conduct a non-traditional Pilates session. This is because stretching exercises will be excluded. The muscle strengthening exercises will be the same as in the TP group, so that it is possible to discuss the influence of the inclusion/exclusion of stretching for the considered outcomes. The total duration of the intervention in this group should be approximately 35 minutes.
  Arms: Pilates without stretching

SUMMARY:
Introduction: The practice of stretching is commonly used in the preparation of activities and/or physical exercises that require some component of flexibility, strength, endurance and muscle power. This explains the high growth in recent decades of studies investigating the effect of stretching, mainly static and dynamic, when performed immediately before activities that aim to develop these physical capacities. Despite the growing interest of scholars on this topic, the long-term impact of dynamic stretching on flexibility, strength performance, endurance and muscle power is still not fully understood. In addition, a type of dynamic stretching little explored in the literature needs investigation: the stretches used during Pilates exercise sessions. The effects of these stretching exercises on a physical conditioning program based on Pilates exercises in the young adult population are not yet known. Objective: To verify through a randomized clinical trial the effects of stretching in a conditioning program based on Pilates exercises on flexibility, strength, endurance and muscle power. Methods: In this study, 32 young adults of both sexes will be randomized into two groups: 1) Traditional Pilates; 2) Pilates Without Stretching. The Traditional Pilates group will perform a protocol of stretching exercises followed by muscle strengthening. The Pilates Without Stretching group will perform an exercise protocol consisting only of muscle strengthening exercises. Muscle strength results will be evaluated by 1 repetition max by elastic resistance; trunk muscle strength/endurance by the 1-minute abdominal test and the Sorensen test, respectively; vertical jump performance by the sargent jump test; handgrip strength by the handheld dynamometer and flexibility by the sit-and-reach test. These physical capacities will be assessed at baseline and after 8 weeks of intervention. Interventions will be performed three times a week for 8 weeks. The analysis will be performed with intent-to-treat analysis and adjusted covariance for baseline outcomes.

ELIGIBILITY:
Inclusion Criteria:

* women between 18 and 45 years of age
* normoweights (Body mass index between 21 to 25 kg/m2)
* not be participating in physical exercise programs for at least six months
* be healthy, according to the Physical Activity Readiness Questionnaire
* not report any medical restrictions for physical exercise
* no history of injury, trauma or illness within the last six months
* not having undergone previous surgery in the last six months
* not have musculoskeletal, cardiorespiratory and neurological disorders that prevent the performance of assessment and intervention protocols
* not be under the action of medications that cause muscle relaxation or that can inhibit muscle tonic action
* not use food supplements or anabolic steroids
* not being on a calorie-restricted diet

Exclusion Criteria:

* start practicing another type of physical exercise during the study period
* not being able to perform the pre-intervention assessment or the intervention exercise protocol
* emergence of lesions that do not allow the continuity of interventions
* withdraw from participating in the study

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2022-09-05 (Actual); Primary Completion 2022-11-25 (Actual); Study Completion 2022-11-25 (Actual)

PRIMARY OUTCOMES:
Change in muscle strength of knee extensors | Pre (baseline) and post-intervention assessment (after 8-weeks)
  Assessment of muscle strength with elastic resistance
Change in strength/endurance by 1-minute sit-up test | Pre (baseline) and post-intervention assessment (after 8-weeks)
  Assessment of abdominal muscle strength/endurance in 1-minute
Change in muscle strength by handgrip test using hand dynamometer | Pre (baseline) and post-intervention assessment (after 8-weeks)
  Assessment of handgrip muscle strength
Change in the muscular resistance of the trunk extensors by the Sorensen test | Pre (baseline) and post-intervention assessment (after 8-weeks)
  Assessment of the muscular resistance of the trunk extensors (Sorensen)

SECONDARY OUTCOMES:
Lower limb muscle power | Pre (baseline) and post-intervention assessment (after 8-weeks)
  Assessment of lower limb muscle power by vertical jump
Flexibility | Pre (baseline) and post-intervention assessment (after 8-weeks)
  Flexibility assessment by the sit-and-reach test

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade Estadual do Norte do Paraná, Jacarezinho, Paraná, Brazil

IPD SHARING:
Plan to Share IPD: No
Data regarding the study will be shared in the publication linked to this record, as a main part of the manuscript and supplementary documents when necessary.

REFERENCES:
- [Derived] Dos Reis AL, de Oliveira LC, de Oliveira RG. Effects of stretching in a pilates program on musculoskeletal fitness: a randomized clinical trial. BMC Sports Sci Med Rehabil. 2024 Jan 8;16(1):11. doi: 10.1186/s13102-024-00808-6. PMID 38191589